CLINICAL TRIAL: NCT05006183
Title: Characterization of Coronary Artery Hemodynamic Measurements and Virtual Angioplasty Planning by Instantaneous Wave-free Ratio (iFR) in Multivessel Acute Coronary Syndrome Patients With Evaluation of the Impact on Clinical Outcomes.
Brief Title: Instantaneous Wave-free Ratio Guidance Strategy Evaluation in the Treatment of Multivessel Acute Coronary Syndrome.
Acronym: iStrategy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daugavpils Regional Hospital (Other Government)
Collaborators: Riga Stradins University (Other)
Responsible Party: Principal Investigator, Deniss Vasiljevs, Principal Investigator, Daugavpils Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0001
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Ischemia; Acute Coronary Syndrome
Keywords: iFR; Instantaneous wave free ratio; virtual percutaneous coronary intervention; Acute coronary syndrome; Multivessel
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iFR-guided (Experimental): One-stage, virtually planned, iFR-guided and optimized PCI.
  Interventions: Procedure: PCI
- Angiography-guided (Active Comparator): Standard practice staged angiography-guided PCI
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — Percutaneous coronary intervention with Drug-Eluting Stents

SUMMARY:
A single-center, prospective, randomized, open-label, blinded end-point clinical trial of instantaneous wave-free ratio (iFR) guidance strategy impact on clinical outcomes in multivessel acute coronary syndrome (ACS) patients.

DETAILED DESCRIPTION:
The "all-comers" study population consists of hemodynamically stable de novo ACS patients with a stenosis of 50% and more by visual estimation in at least two separate coronary arteries with Thrombolysis in Myocardial Infarction (TIMI) flow ≥ 2 and willing to sign a patient informed consent. ACS diagnosis established by angina pectoris symptoms and/or ECG changes and/or hs-troponin I levels. The use of drug-eluting stents is mandatory in both treatment groups. In the intervention strategy group, patients are treated by the iFR-guided percutaneous coronary intervention (PCI) in one stage. In the control group, patients are treated in accordance with the standard practice of angiography-guided staged approach.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* willing to give informed consent
* hemodynamically stable de novo acute coronary syndrome patients with a stenosis of 50% and more by visual estimation in at least two separate coronary arteries
* adequate coronary flow, Thrombolysis in Myocardial Infarction (TIMI) flow ≥ 2
* sinus rhythm

Exclusion Criteria:

* inability to give consent;
* younger than 18 years of age
* atrial fibrillation rhythm at the time of inclusion
* with significant valve disease
* in cardiogenic shock
* with reduced kidney function - eGFR < 30 (mL/min/1.73m2);
* with congenital heart defects
* with acute pulmonary artery embolism;
* with isolated left main ostial stenosis;
* on active oncologic treatment or toxic cardiomyopathy;
* revascularization by PCI is not possible due to other comorbidities or patient denial of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
PCI-related Major adverse cardiac events (MACE) | Index admission
  Composite of cardiac death, non-fatal myocardial infarction, unplanned revascularization, stent thrombosis, flow limiting coronary dissections, no-reflow phenomenon, coronary perforations, coronary distal embolization, vascular access site complications requiring blood transfusion or surgical intervention and contrast-induced nephropathy requiring hospitalisation.
PCI-related Major adverse cardiac events (MACE) | 3 months
  Composite of cardiac death, non-fatal myocardial infarction, unplanned revascularization, stent thrombosis, flow limiting coronary dissections, no-reflow phenomenon, coronary perforations, coronary distal embolization, vascular access site complications requiring blood transfusion or surgical intervention and contrast-induced nephropathy requiring hospitalisation.
PCI-related Major adverse cardiac events (MACE) | 12 months
  Composite of cardiac death, non-fatal myocardial infarction, unplanned revascularization, stent thrombosis, flow limiting coronary dissections, no-reflow phenomenon, coronary perforations, coronary distal embolization, vascular access site complications requiring blood transfusion or surgical intervention and contrast-induced nephropathy requiring hospitalisation.

SECONDARY OUTCOMES:
Segmental myocardial deformation by speckle-tracking echocardiography | Index admission, 3 months and 12 months
  Change of segmental myocardial deformation
Health-related Quality of Life | Index admission, 3 months and 12 months
  Change in health-related quality of life measured using the EQ-5D-5L questionnaire
Number of Participants with Decline of eGFR | Index admission, 3 months and 12 months
  Number of participants with decline of eGFR 30% and more in comparison to the first eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Deniss Vasiljevs, MD, Principal Investigator — Daugavpils Regional Hospital
Locations (1):
- Daugavpils Regional Hospital, Daugavpils, Latvia

IPD SHARING:
Plan to Share IPD: No